CLINICAL TRIAL: NCT00710827
Title: A 54 Week Treatment, Randomized, Multi Center, Double Blind, Placebo Controlled Study to Assess the Safety and Efficacy of NEBIDO 1000 mg (4 ml) in Elderly Men With Symptomatic Late Onset Hypogonadism (SLOH)
Brief Title: Nebido Versus Placebo in Elderly Men With Typical Symptoms of Late Onset Hypogonadism Over a Period of 54 Weeks
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91579; 2008-002053-20 (EudraCT Number); 310874 (Other: company internal)
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Hypogonadism
Keywords: NEBIDO,; Hypogonadism,; Symptomatic late onset,; Testosterone deficiency
MeSH Terms: conditions — Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: NEBIDO
- Arm 2 (Placebo Comparator)
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: NEBIDO — Patients will receive 54 weeks of treatment with Nebido, 5 intramuscular injections of 4ml Nebido (at baseline, week 6, 18, 30, 42)
  Arms: Arm 1
Drug: PLACEBO — Patients will receive 54 weeks of treatment with placebo, 5 intramuscular injections of 4ml placebo (at baseline, week 6, 18, 30, 42)
  Arms: Arm 2

SUMMARY:
To evaluate the safety and efficacy of Nebido compared to placebo in elderly men aged 50 and over with symptomatic late onset hypogonadism

DETAILED DESCRIPTION:
Explorative objectives: Change in grip strength (Subgroup only: optional for sites with experienced in testing muscle function); Change in physical performance test i.e. lower limb muscle strength (subgroup only; optional for sites experienced in testing muscle function). Please note that the 2 explorative objectives mentioned above must be performed together. All measured at baseline, week 30, week 54, no safety measure. Safety parameters Prostate safety: digital rectal examination (DRE) Measured at screening, week 30+ 54, safety measure. International prostate symptom score (IPSS): International prostate symptom score (IPSS) Measured at screening, week 18, 30, 42, 54, safety measure. Laboratory tests for lipids (total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides) and liver function tests (aspartate aminotransferase (AST) and alanine transaminase (ALT)) Measured at screening, week 6, 18, 30, 42, 54, safety measure. Standard laboratory tests for androgen treatment: prostate specific antigen (PSA); hemoglobin; hematocritMeasured at screening, week 6, 18, 30, 42, 54, safety measureAdverse eventsMeasured at screening, baseline, week 6, 18, 30, 42, 54Vital signsMeasured at screening, week 18, 30, 42, 54, safety measure.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 50 years and older
* Symptomatic hypogonadism as defined by a) and b):
* a) Total testosterone below 12nmol/l
* b) Aging males symptom score above 36
* Willing to avoid significant change in the pattern of physical exercise and lifestyle for the duration of the study
* Willing to voluntarily sign a statement of informed consent to participate in the study.

Exclusion Criteria:

* Use of androgen therapy or anabolic steroids
* Suspicion or known history of liver tumors, prostate or breast cancer
* Hypersensitivity to the active substances or any of the excipients of NEBIDO e.g. Benzyl benzoate and castor oil. Hypercalcemia accompanying malignant tumors
* Blood coagulation irregularities presenting an increased risk of bleeding after intramuscular injections sleep apnea
* Polycythemia
* Hematocrit level >50% at entry to the study (i.e. screening visit/visit 1)
* Patients using 5-a-reductase inhibitors such as finasteride or dutasteride should be excluded from the study.
* Prolactin level >25ng/ml
* Organic hypothalamic-pituitary pathology
* Prostate specific antigen (PSA) level ≥ 4ng/ml
* Severe symptomatic benign prostatic hyperplasia (IPSS sum score ≥ 20)
* Epilepsy not adequately controlled by treatment
* Migraine not adequately controlled by treatment
* Patients requiring or undergoing fertility treatment
* Any clinically significant chronic disease that might, in the opinion of the investigator, compromise patient's safety interfere with the evaluations, or preclude completion of the trial (e.g. hemochromatosis, chronic lung disease, chronic malabsorption disease)
* Known history of alcohol or drug abuse
* Medical, psychiatric or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol, or to complete the study.
* Hypertension which is not adequately controlled on therapy
* Severe cardiac, hepatic or renal insufficiency
* Coronary heart disease not stabilized by therapy as assessed by the investigator
* Metal implants in the body (metal implants in the head will not exclude patients from participation)
* Concomitant participation in another clinical trial within 1 month of entry into this study (i.e. randomized and has taken study medication).

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
To assess the change from baseline in lean body mass after 54 weeks of treatment with NEBIDO compared to placebo | Baseline, week 30, week 54

SECONDARY OUTCOMES:
Change from baseline in total body mass | Baseline, week 30, week 54
Change from baseline in fat mass | Baseline, week 30, week 54
Change from baseline in bone mineral density | Baseline, week 30, week 54
Aging Male Symptoms (AMS) rating scale | Baseline, week 30, week 54
International Index of Erectile Function- erectile function domain (IIEF-EF) | Baseline, week 30, week 54
Change in serum levels of testosterone (central laboratory) | Baseline, week 30, week 54
Change in waist circumference | Baseline, week 30, week 54

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- Germany (2):
  - Bonn, North Rhine-Westphalia
  - Halle, Saxony-Anhalt
- Italy (3):
  - Milan
  - Napoli
  - Roma
- Riga, Latvia
- Poland (3):
  - Lodz
  - Warsaw
  - Wroclaw
- Russia (4):
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Volgograd
- United Kingdom (8):
  - Reading, Berkshire
  - London, London
  - Manchester, Manchester
  - Lichfield, Staffordshire
  - Glasgow, Stratchclyde
  - Birmingham, West Midlands
  - Cardiff
  - Chorley